CLINICAL TRIAL: NCT05676580
Title: Risk Factors and Progression of Keratoconus
Acronym: FRPK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RECHMPL20_0450 / UF8090
Record Dates: First submitted 2022-12-18; First posted 2023-01-09 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abstention (Other): After keratoconus diagnosis the patient won't be assigned to intervention
  Interventions: Other: abstention
- Intervention (cross-linking surgery or intra corneal ring) (Other): After keratoconus diagnosis the patient was assigned to cross linking surgery or intra corneal ring surgery
  Interventions: Procedure: cross-linking surgery or intra corneal ring

INTERVENTIONS:
Procedure: cross-linking surgery or intra corneal ring — After keratoconus diagnosis the patient was assigned to surgery
  Arms: Intervention (cross-linking surgery or intra corneal ring)
Other: abstention — No surgery
  Arms: Abstention

SUMMARY:
Primary objective :

Description of keratoconus at baseline and during progression in 200 participants followed by the ophthalmology departments of CHU Montpellier, CHU Bordeaux and CHU Toulouse during a 2-year period. Clinical outcome, histology of the cornea and tears proteomics will be assessed in 4 groups at different points in time:

* At 6 months in participants with no intervention (risk reduction instructions: not to rub their eyes)
* At 6 months in participants with no intervention that didn't comply with the risk reduction instructions
* At 1 month in participants assigned to cross-linking surgery
* At 1 month in participants assigned to intra corneal ring surgery If both eyes are affected, both will be evaluated with their own visit agenda. Visits for no surgery participants will be set at 6 months, 12 months and 24 months in the absence of intervention (apart from the behavioral risk reduction).

Visits for surgery participants will be set at D7, 1 month, 6 months, 12 months and 24 months after the procedure: cross-linking or placement of the intra corneal ring.

Secondary objective :

Description of the association between clinical outcomes, histological progression of the cornea and tears proteomics in time, 2 years period.

Comparison of tears proteomics in 36 participants with keratoconus followed at CHU of Montpellier and healthy participants at baseline .

DETAILED DESCRIPTION:
This trial is a prospective cohort study of 200 participants with keratoconus followed by the ophthalmology departments of CHU Montpellier, CHU Bordeaux and CHU Toulouse during a 2-year period. If both eyes are affected, each will be evaluated considering their own visit agenda. Histological and proteomic evaluations will be performed in 36 participants's eyes whose initial management is abstention of surgery (12 participants), cross-linking (12 participants) or intra corneal ring (12 participants).

The target population consist of participants with clinical keratoconus (topographic Rabinowitz criteria with slit lamp abnormalities and visual impairment), preclinical or crude keratoconus (abnormal or suspicious topography with normal slit lamp examination and normal visual acuity). They will be aged between 10 and 40 years included.

The follow-up will be taken care off by the ophthalmology departments of the Montpellier University Hospital, Bordeaux University Hospital or Toulouse University Hospital Collection of written informed consent, after a period of reflection, will be necessary for adult participants. For minors: informed consent will have to be signed by at least one of the 2 parents or legal guardians, and approval from the child will be asked after a period of reflection. All participants will have to be affiliated to the French social security system or beneficiary of such a system.

Description of the study course:

No therapeutic intervention outside of routine care will be performed. Depending on the therapeutic orientation, the follow-up is carried out as follows:

* Visits at 6 months, 12 months and 24 months in the absence of intervention (apart from the behavioral risk reduction management).
* Visits at day 7, 1 month, 6 months, 12 months and 24 months after the procedure: cross-linking or placement of the intra corneal ring.

In this study, participants will be followed for a maximum of 2.5 years. In addition to the description of keratoconus progression, we will take a tear sample using the Schirmer test to create a biobank. This tears collection will be performed in 36 participants followed at the Montpellier University Hospital, at inclusion and at short-term follow-up visit (6 months if abstention, 1 month if surgery).

Judging criteria:

* Paraclinical examination of the participants
* Ophthalmological paraclinical data
* Confocal microscopy examination
* ABCD classification of keratoconus
* Composition and evolution of tears determined by proteomic analysis
* Survey on risk factors: allergies, atopy, ocular friction, family history, ethnic origin, smoking, dry eye syndrome, low pachymetry

Prevalence of risk factors: a survey will measure the prevalence of risk factors for keratoconus:

* Presence of atopy/allergy
* Eye rubs
* Family history
* Ethnic origin
* Tobacco use
* Dry eye syndrome (survey + clinical examination)
* Low pachymetry

This self-survey will be completed at the inclusion visit and at the last follow-up visit (M24). The time to complete this questionnaire is approximately 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Participants with clinical keratoconus (Rabinowitz criteria with topographic slit lamp abnormalities and visual impairment), preclinical or crude keratoconus (abnormal or suspicious topography with normal slit lamp examination and normal visual acuity, visual acuity)
* Followed by the ophthalmology services of the CHU Montpellier, CHU Bordeaux or CHU Toulouse
* For adult Participants: collection of written informed consent, after a period of reflection period
* For minors: informed consent signed by at least one of the 2 parents or legal representatives legal representatives, and assent of the child after a period of reflection
* Affiliation to the French social security system or beneficiary of such a system

Exclusion Criteria:

* Person under legal supervision, guardianship or curator
* History of corneal implant on both eyes
* Planned relocation before the end of the first stage of treatment (abstention, cross-linking, intra-corneal ring depending on the participant)

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2027-06-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Keratoconus clinical progression (Keratometry map) | Baseline vs Visit at 1 month/6 months/12 months/24 months
  Modelisation of refraction measurements in diopters, by corneal elevation topography (Orbscan and Pentacam), giving an additional indicator of the corneal deformity. High values of diopter correspond to positive bulges of the cornea. A topographic axial map will be acquired to monitor minimal and maximal keratometry.
  These measurements will be taken at baseline and compared for reference of progression at each visit for each eye.
  Keratoconus definition according to Rabinowitz (Rabinowitz YS, 1989) criteria:
  * Corneal asymmetry greater than 1.5 diopters (D), between the upper and lower part of the cornea, on the median vertical axis.
  * Central corneal power (Kmax) > 47.2 D, measured at the top of the cone.
  * Asymmetry of central keratometry > 1D between the two eyes
Keratoconus clinical progression (Pachymetric map) | Baseline vs Visit at 1 month/6 months/12 months/24 months
  Thickness of the cornea will be assessed in microns (µm) at several locations and will be presented as a map by corneal elevation topography (Orbscan and Pentacam).
  The pachymetric map will be acquired at baseline and compared for reference of progression at each visit for each eye. The higher and lower thickness points will be notified for the anterior and posterior parts of the eye.
Keratoconus clinical progression (Visual acuity test) | Baseline vs Visit at 1 month/6 months/12 months/24 months
  Visual acuity test with and without correction: decimal and Parinaud scales secondarily translated in LogMar.
Keratoconus clinical progression (Biomicroscopic examination of the cornea) | Baseline vs Visit at 1 month/6 months/12 months/24 months
  A biomicroscopic examination of the cornea in search of signs that may modify the therapeutic indications i.e : Fleischer rings (iron deposits in the lower part of the bulge, due to the stagnation of tears), visible corneal nerves, corneal opacities (due to scar tissue)
ABCD grading of keratoconus | Baseline vs Visit at 1 month/6 months/12 months/24 months
  Grading of the keratoconus, according to the ABCD classification :
  * A: keratometry of the anterior surface of the cornea (Anterior radius of curvature (ARC)), in the area of 3 mm centered by the thinnest point.
  * B: keratometry of the posterior surface of the cornea (Back or posterior radius of curvature PRC), in the 3mm area centered by the thinnest point.
  * C: thinnest point of the Cornea, i.e. minimum pachymetry.
  * D: Distance best corrected vision: visual acuity with the best correction, measured in 10° or in the Parinaud scale.
Keratoconus histological progression - Confocal microscopy (tissue thickness) | Baseline vs Visit at 1 month/6 months/12 months/24 months
  Histological degradation of the cornea taken at baseline for reference. The confocal microscope allows longitudinal analysis making it possible to carry out comparative qualitative and quantitative analyzes of the corneal tissue during time. In keratoconus, this technique is possible to highlight a reduction in basal plexus nerve density and poorer anterior stromal cell density compared to healthy subjects.
  Tissue thickness in microns (µm)
Keratoconus histological progression - Confocal microscopy (Cellular organization) | Baseline vs Visit at 1 month/6 months/12 months/24 months
  Histological degradation of the cornea taken at baseline for reference. The confocal microscope allows longitudinal analysis making it possible to carry out comparative qualitative and quantitative analyzes of the corneal tissue during time. In keratoconus, this technique is possible to highlight a reduction in basal plexus nerve density and poorer anterior stromal cell density compared to healthy subjects.
  Cell organization and morphology. Image acquisition.
  * Colonization by inflammatory cells (yes/no), increased nucleo/cytoplasmic ratio (yes/no), hyperreflectivity of the nuclei (yes/no).
  * Nerve density of the basal plexuses of normal appearance (yes/no), straight with branches (yes/no), normal hyperreflectivity (yes/no)
Keratoconus histological progression - Confocal microscopy (Cellular density) | Baseline vs Visit at 1 month/6 months/12 months/24 months
  Histological degradation of the cornea taken at baseline for reference. The confocal microscope allows longitudinal analysis making it possible to carry out comparative qualitative and quantitative analyzes of the corneal tissue during time. In keratoconus, this technique is possible to highlight a reduction in basal plexus nerve density and poorer anterior stromal cell density compared to healthy subjects.
  Cellular density (number). Image acquisition.
  - Cell count in the different layers, corneal nerve count from the basal plexus to the corneal apex
Keratoconus histological progression - Confocal microscopy (Light scattering) | Baseline vs Visit at 1 month/6 months/12 months/24 months
  Histological degradation of the cornea taken at baseline for reference. The confocal microscope allows longitudinal analysis making it possible to carry out comparative qualitative and quantitative analyzes of the corneal tissue during time. In keratoconus, this technique is possible to highlight a reduction in basal plexus nerve density and poorer anterior stromal cell density compared to healthy subjects.
  Light scattering in vivo, measurement of corneal deformity. Diopter.
Risk factors - Questionnaire | Baseline vs 24 months
  * Presence of atopy/allergy
  * Eye rubbing
  * Family medical history
  * Ethnicity
  * Smoking habits
  * Dry eye syndrome
Tears proteomics | Baseline vs Visit at 1 month/6 months
  For 36 participants from Montpellier. Composition and evolution of tears determined by proteomic analysis

SECONDARY OUTCOMES:
ABCD class worsening between consultations | Baseline vs Visit at 1 month/6 months - Baseline vs 12 months - Baseline vs 24 months
  At baseline and during follow-up
Keratoconus histological evolution | Baseline vs Visit at 1 month/6 months
  Comparison of confocal microscopy results from primary outcomes through time.
Proteomic profile evolution | Baseline vs Visit at 1 month/6 months
  Difference between the composition of tears from healthy participants and from keratoconus patients from baseline to short term follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent DAIEN, PR, Principal Investigator — CHU Monptellier
Locations (1):
- CHU Gui de Chauliac - Service d'Ophtamologie, Montpellier, Occitanie, France

IPD SHARING:
Plan to Share IPD: Undecided